CLINICAL TRIAL: NCT02068911
Title: Validation of the Measure of ETCO2, Compared to PTCO2 and PaCO2 in the Home-ventilated Neuromuscular Patient
Brief Title: Concordance Between ETCO2, PTCO2 and PaCO2 in the Home-ventilated Neuromuscular Patient
Acronym: Capnovivo
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A01629-36
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Neuromuscular Disease; Chronic Respiratory Insufficiency; Intermittent Positive-pressure Ventilation
Keywords: Neuromuscular disease; Home ventilation; End tidal CO2; Transcutaneous CO2; Monitoring
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Monitoring of ETCO2 and PTCO2: All neuromuscular patients
  Interventions: Device: Monitoring of ETCO2 and PTCO2

INTERVENTIONS:
Device: Monitoring of ETCO2 and PTCO2 — Concomitant monitoring of ETCO2 and PTCO2
  Other Names: PTCO2: Sentec Capno-Oxymetry (Sentec); ETCO2: Module of the BREAS Vivo 50 home ventilator

SUMMARY:
The purpose of this study is to compare the measure of the CO2 obtained on the end-tidal expiratory gas (ETCO2) with the value of CO2 obtained by transcutaneous measure (PTCO2), in home-ventilated neuromuscular patients.

DETAILED DESCRIPTION:
Monitoring of the effectiveness of ventilation in patients with neuromuscular require to regularly measure blood gases and in particular carbon dioxide (CO2). The reference technique is arterial puncture. In recent years, a non-invasive techniques measuring CO2 by transcutaneous sensor (PTCO2) was introduced among the tools regularly used for follow-up monitoring of home ventilated patients.

Another technique for monitoring CO2, originally developed for anesthesia, is based on the measurement of exhaled CO2 (ETCO2). This technique requires relatively simple equipment, and represents a potential alternative for monitoring home-ventilated patients.

Recently, sensors for ETCO2 were coupled to devices for home ventilation. To the best of our knowledge, the role of ETCO2 in monitoring long-term ventilated patients has not been investigated to date.

The purpose of the study is to analyze the correlation between the two non-invasive methods for measuring CO2: PTCO2 and ETCO2, in a group of home-ventilated patients with neuromuscular disease.

The patients will be recruited during a routine follow-up hospitalization for their home-ventilation, and the ETCO2 will be measured during one night, in addition to the routinely measured PTCO2.

ELIGIBILITY:
Inclusion Criteria:

* Patient with neuromuscular disease, treated with home invasive or non-invasive ventilation
* Male or female age higher or equal to 18 years
* Negative pregnancy test for women of childbearing age or having an effective contraception

Exclusion Criteria:

* Acute Respiratory Failure
* Long-term oxygen therapy
* Refusal to participate in the study
* Plan of legal protection
* Pregnant Women
* Failure to cooperate
* No affiliation to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited among the neuromuscular patients treated at the University Hospital Raymond Pointcaré, Garches (France), during a routine follow-up hospitalization for their home-ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
concordance between the nocturnal average values of ETCO2 and PTCO2 | one night
  concordance between the nocturnal average values of the CO2 measured by the two non-invasive techniques ETCO2 and PTCO2

SECONDARY OUTCOMES:
concordance between the nocturnal maximal values of ETCO2 and PTCO2 | one night
  concordance between the nocturnal maximal values of the CO2 measured by the two non-invasive techniques ETCO2 and PTCO2
concordance between the variation of the values of ETCO2 and PTCO2 | one night
  concordance between the variation of the values of the CO2 measured by the two non-invasive techniques ETCO2 and PTCO2
concordance between the values of ETCO2, PTCO2 and arterial CO2 (PaCO2) measured at the same time | one night
  concordance between the values of ETCO2, PTCO2 and arterial CO2 (PaCO2) measured at the same time

OTHER OUTCOMES:
influence of circuit leakage on the gradient between PaCO2 and ETCO2 | one night
  evaluate the influence of circuit leakage on the gradient between PaCO2 and ETCO2

CONTACTS AND LOCATIONS:
Overall Officials: Adam OGNA, MD, Principal Investigator — HOPITAL RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France

REFERENCES:
- [Derived] Orlikowski D, Prigent H, Ambrosi X, Vaugier I, Pottier S, Annane D, Lofaso F, Ogna A. Comparison of ventilator-integrated end-tidal CO2 and transcutaneous CO2 monitoring in home-ventilated neuromuscular patients. Respir Med. 2016 Aug;117:7-13. doi: 10.1016/j.rmed.2016.05.022. Epub 2016 May 24. PMID 27492508